CLINICAL TRIAL: NCT01392027
Title: Biospecimens for the Early Detection, Prevention, Diagnosis and Treatment of Diseases of the Pancreas.
Brief Title: Biospecimens for Identification of Diseases of the Pancreas.
Acronym: SPORE-PANC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Missy Tuck, Project manager, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: P50-CA13081001A2
Record Dates: First submitted 2011-07-06; First posted 2011-07-12 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Pancreatic Cancer; Chronic Pancreatitis; Type II Diabetes; Pancreatic Cysts; Healthy Control
Keywords: Pancreatic Cancer; Chronic Pancreatitis; Diseases of the pancreas
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatitis, Chronic; Diabetes Mellitus, Type 2; Pancreatic Cyst; Pancreatic Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Blood Draw — Blood draw for research specimens only

SUMMARY:
This proposed project is designed to collect data and specimens from patients/subjects presenting to the University of Michigan with a disease affecting the pancreas (or specific control populations). This protocol is focused on collecting data, blood samples, and tissue on subjects with pancreatic diseases, including pancreatic cancer, pancreatic cysts, pancreatitis, diabetic controls, jaundice/biliary obstruction controls, and otherwise healthy controls.

We are collecting up to 50 mls of blood for research purposes only. Plasma, serum and buffy coat are collected and stored according to strict SOPs.

DETAILED DESCRIPTION:
The recently funded GI SPORE, here at the University of Michigan, is focused on pancreatic and colon diseases. This protocol is focused on collecting data, blood samples, and tissue on subjects with pancreatic diseases, including pancreatic cancer, pancreatic cysts, pancreatitis, diabetic controls, jaundice/biliary obstruction controls, and otherwise healthy controls. A SPORE is an NCI-funded, Specialized Program in Research Excellence, with specific requirements. Those requirements include 4 projects with a clinical and a basic science Co-PI and several COREs, including a biospecimen core. Each project that has a human subjects component will require a separate protocol and IRB submission when those projects are to begin.

The specific populations we are recruiting are determined by the aims of project 2 and by the need to create a repository as part of the biospecimen core (please see the grant for details on the aims of these 2 projects).

A specially designed database is being built for this study to handle the data aspects. Our collaborators at Dartmouth College have significant experience in managing data as they have been our partners for our work in the EDRN (PI Brenner). Case report forms and other data collection tools have been developed and are being used to populate the database. All of the actual data will be completely deidentified per HIPAA regulations.

We intend to model the data and specimen collection on the model used by our work with the NCI-EDRN. This includes a customized database, the use of kits with pre-labled, bar-coded aliquots, and standardized data collection forms (CRFs).

ELIGIBILITY:
Inclusion Criteria:

Overall Inclusion (all subjects must meet these criteria to be enrolled)

* Adults 18 years of age or older
* Able to physically tolerate removal of 50 ml of blood
* Willing to sign informed consent.

Exclusion Criteria:Overall Exclusion (for all subjects)

* Pregnant or lactating
* Known HIV/AIDS or Hepatitis C
* Prepped for colonoscopy at the time of blood collection
* Unable to understand English
* Receiving chemotherapy or radiation at time of enrollment
* Any cancer within 5 years of enrollment except any of the following:

  * Squamous cell carcinoma of the skin or Basal cell carcinoma of the skin
  * Carcinoma in situ of the cervix, Stages Ia or Ib invasive squamous cell carcinoma of the cervix treated by surgery only. (Excluded if had pelvic radiation)
  * Stage Ia Grade 1 adenocarcinoma of the endometrium treated with surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 712 (Actual)
Dates: Start 2011-04; Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Validation of glycoprotein panel as a pancreatic cancer biomarker | 5 years
  To create a set of cases and controls to validate a novel glycoprotein panel for non-invasive or early detection of pancreatic cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- Univerisity of Michigan, Ann Arbor, Michigan, United States